CLINICAL TRIAL: NCT06814808
Title: Comparison of Three Different Myofascial Trigger Point Treatments on Pain, Range of Motion, Joint Position Sense and Quality of Life in Chronic Non-specific Neck Pain
Brief Title: Comparison of Three Different Myofascial Trigger Point Treatments in Chronic Non-Specific Neck Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BiruniUni.
Record Dates: First submitted 2025-01-02; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Chronic Non-specific Neck Pain
Keywords: Strain Counterstrain; Integrated Neuromuscular Inhibition Technique; Ischaemic compression; Chronic non-specific neck pain; Manual therapy; Exercise; Conventional physiotherapy programme
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ischaemic Compression Group (Active Comparator): Ischaemic compression Manual therapy
  Interventions: Other: Conventional Therapy; Other: Ischemic Compression Group
- Strain Counterstrain Group (Experimental): Strain Counterstrain Manual therapy
  Interventions: Other: Conventional Therapy; Other: Strain-Counter Strain
- Integrated Neuromuscular Inhibition Technique Group (Experimental): Integrated Neuromuscular Inhibition Technique Manual therapy
  Interventions: Other: Conventional Therapy; Other: Integrated Neuromuscular Inhibition Technique (INIT)

INTERVENTIONS:
Other: Conventional Therapy — All three groups will receive a conventional physiotherapy program (TENS, therapeutic ultrasound, hot pack) 5 times a week for 4 weeks and the same exercise program 3 days a week for 4 weeks.
Other: Ischemic Compression Group — The ischemic compression group will receive ischemic compression therapy for the upper trapezius, levator scapulae, splenius capitis, and lower trapezius muscles.
  Arms: Ischaemic Compression Group
Other: Strain-Counter Strain — The strain counterstrain technique will be applied to the upper trapezius, levator scapulae, splenius capitis, and lower trapezius muscles.
  Arms: Strain Counterstrain Group
Other: Integrated Neuromuscular Inhibition Technique (INIT) — This group will be subjected to INIT for the upper trapezius, levator scapulae, splenius capitis, and lower trapezius muscles, 3 sessions per week for 4 weeks (12 sessions in total).
  Arms: Integrated Neuromuscular Inhibition Technique Group

SUMMARY:
The aim of this study was to compare the efficacy of ischaemic compression (IC), positional relaxation (Strain Counterstrain [SCS]), and integrated neuromuscular inhibition technique (INIT) applications on pain intensity, pressure pain threshold, range of motion, joint position sense, disability, kinesiophobia, quality of life and patient satisfaction in addition to conventional treatment for chronic non-specific neck pain.

It is planned to include 51 patients in the study. The included patients will be divided into 3 groups: Group 1 (HR Group), Group 2 (SCS Group) and Group 3 (INIT Group). All three groups will receive a conventional physiotherapy programme 5 times a week for 4 weeks and the same exercise programme 3 days a week for 4 weeks.

DETAILED DESCRIPTION:
Chronic neck pain is one of the most common musculoskeletal problems in the general population and is the second most common type of pain after low back pain worldwide. Electrophysiological agents, therapeutic exercise and trigger point therapy techniques are frequently used in chronic non-specific neck pain. There is insufficient evidence in the current literature regarding which trigger point therapy technique is more effective. The aim of this study was to compare the efficacy of ischaemic compression (IC), positional relaxation (Strain Counterstrain [SCS]), and integrated neuromuscular inhibition technique (INIT) on pain intensity, pressure pain threshold, range of motion, joint position sense, disability, kinesiophobia, quality of life and patient satisfaction in addition to conventional treatment for chronic non-specific neck pain. The study was planned to include 51 patients between the ages of 18-65 years who applied to Gebze Medicalpark Hospital and met the inclusion criteria. The included patients will be randomised and divided into 3 groups: Group 1 (HR Group), Group 2 (SCS Group) and Group 3 (INIT Group). All three groups will receive a conventional physiotherapy programme (TENS, therapeutic ultrasound, hot pack) 5 times a week for 4 weeks and the same exercise programme 3 days a week for 4 weeks. In addition to conventional treatment, Group 1 will receive HR for upper trapezius, levator scapulae, splenius capitus and lower trapezius muscles, Group 2 will receive SCS for upper trapezius, levator scapulae, splenius capitus and lower trapezius muscles and Group 3 will receive INIT for upper trapezius, levator scapulae, splenius capitus and lower trapezius muscles 3 sessions per week for 4 weeks (12 sessions in total). As evaluation criteria, visual analogue scale will be used to evaluate the intensity of pain felt at rest, activity and at night, and algometer will be used to objectively measure pain threshold and tolerance. Cervical range of motion and joint position sense will be assessed using CROM III-Cervical Range of Motion device. Disability level will be assessed using the Neck Disability Scale, fear of movement using the Tampa Kinesiophobia Scale, quality of life using the Short Form-12, and Global Change Scale to assess patient satisfaction. Assessments will be made before starting the treatment programme and after the completion of the 4-week treatment programme.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between 18 and 65 years of age,
* The patient presents to the outpatient clinic with a complaint of neck pain that has been persisting for at least 3 months,
* Pain intensity higher than 3.5/10 cm according to the Visual Analogue Scale,
* Active trigger point in at least one of the upper trapezius, levator scapulae, splenius capitus, lower trapezius muscles that may cause neck pain,
* Neck Disability Index total score higher than 15,
* Having the ability to read and write in Turkish was determined as the inclusion criteria.

Exclusion Criteria:

* Has had a neck, spine or shoulder injury within the last 6 months,
* The patient has neck pain caused by inflammatory, hormonal, neurological disorders or after trauma,
* Positive radicular findings compatible with nerve root compression, history of spinal fracture, spinal tumours and related malignancies, congenital spinal anomalies,
* History of neck, upper thoracic spine and shoulder surgery,
* Scoliosis surgery or a health problem that causes limitation in spinal mobility,
* Diagnosed with any malignant condition, systemic, neurological or rheumatological disease,
* Having a skin disease or hearing-vision problem that may affect the assessment process,
* Uncontrolled hypertension, uncontrolled diabetes mellitus, meniere's disease and vertigo,
* Physiotherapy sessions for neck pain in the last month,
* Pregnancy,
* Use of any analgesic or psychotropic agent was determined as exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 weeks
  The intensity of pain felt in the neck area at rest, during activity (cervical flexion, extension, right and left lateral flexion, right and left rotation) and at night will be evaluated numerically using a visual analogue scale (VAS). Individuals will be told that the number '0' on a 10 cm horizontal line indicates 'no pain' and the number '10' indicates 'unbearable pain'. The place marked by the individual will be determined as pain intensity in cm.
Algometer | 4 weeks
  An Algometer (Baseline Push-Pull Force Gauge®, Fabrication Enterprises, Inc.) will be used to objectively measure pain threshold and tolerance. Before measuring with the algometer, a pressure will be applied to the pulp of the thumb of the hand, which is the control point. Then, a force will be applied to the same point to cause pain so that the subject can distinguish between the sensation of pressure and the sensation of pain. Then, at the C2 spine level, the pressure will be applied vertically to the muscle tissue from the midpoint of the right-left paraspinal muscles and the right-left upper trapezius muscles, increasing the pressure by 1kg/cm2 every three seconds until the subject feels pain. The subject will be told to report when he/she feels pain while applying force with the device (kg/ cm²). This process will be repeated three times and the average value will be calculated.
Cervical Joint Position Sense | 4 weeks
  Cervical joint position sense will be evaluated by head repositioning test using CROM III-Cervical Range of Motion (Performance Attainment Associates, Lindstrom, MN) device. The target position will be 25° flexion, extension, right-left lateral flexion, right-left rotation respectively. The subject will sit on a chair with a straight back, knees flexed 90 degrees and feet flat on the floor. The subject will be asked to close his/her eyes. Then, the subject's neck will be passively flexed 25° in a slow rhythm, and the position will be maintained for 5 seconds. The subject will be asked to remember this position. Afterwards, the subject's neck will be passively moved to the neutral position in a slow rhythm. The subject will then be instructed to actively move his/her neck and reposition himself/herself in the target position. The subject will signal by saying 'yes' when repositioned to the target position. The deviation in the repositioning test result will be evaluated as joint positi
Cervical Range of Motion | 4 weeks
  Cervical region flexion-extension, right-left lateral flexion and right-left rotation range of motion will be evaluated using the CROM III-Cervical Range of Motion (Performance Attainment Associates, Lindstrom, MN) device. The device has undergone a reliability study and has been reported as a clinically reliable tool for assessing normal range of motion in the cervical region. The subject will be positioned in an upright sitting position on a chair with back support, with the middle and lower back in contact with the chair, feet on the floor and arms comfortably supported on both sides of the chair. The subject will be asked to look straight ahead. After checking the alignment of the nose, mouth, chin and earlobe and making sure that the cervical region is in the anatomical position, the subject will be commanded to start the movement. Each evaluation will be repeated three times and the average value will be recorded.
Neck Disability Scale | 4 weeks
  It will be evaluated with the Neck Disability Scale. The Neck Disability Scale is based on the Oswestry Low Back Pain Disability Index and consists of 10 items. It includes pain sensitivity, personal care, weight lifting, reading, headaches, concentration, work/study, driving, sleep and social activities. Each question has 6 answer options that measure the severity of pain or limitation. Scoring is done between 0-5. The total score is between 0-50. According to the total score, 0-4 points are classified as no limitation; 5-14 as mild limitation; 15-24 as moderate limitation; 25-34 as severe limitation; 34 and above as completely limited. Turkish validity and reliability study was conducted.
Tampa Kinesiophobia Scale | 4 weeks
  Tampa Kinesiophobia Scale (TKS) will be used. TQS is a scale developed to measure the fear of movement/reinjury. It consists of a total of 17 questions. It includes injury/reinjury and fear-avoidance parameters in work-related activities. It consists of 17 questions in total. Total score varies between 17-68. High scores indicate a high level of kinesiophobia. Turkish validity and reliability study was conducted.
Short Form-12/ SF-12 | 4 weeks
  Short Form-12 (SF-12) will be used to assess quality of life. SF-12 has 2 total measurements including physical (PCS-12) and mental (MCS-12) components, and high scores indicate good health status. This assessment is a shortened version of SF-36. Turkish validity and reliability studies were conducted.
Global Change Scale | 4 weeks
  It will be evaluated using the Global Change Scale (GTS). In order to evaluate the perceived effect of the treatment applied to the patients, it is used to determine the amount of change considering the current health status after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci Olgun, Asst prof., Study Chair — Medeniyet University, Health Sciences Faculty Department; Maryam Zare, MD, Study Chair — Medical Park Gebze; Pınar Atamert, MSc, Principal Investigator — Biruni University, Health Sciences Faculty Department
Locations (1):
- Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

REFERENCES:
- [Background] Dardzinski JA, Ostrov BE, Hamann LS. Myofascial pain unresponsive to standard treatment: successful use of a strain and counterstrain technique with physical therapy. J Clin Rheumatol. 2000 Aug;6(4):169-74. doi: 10.1097/00124743-200008000-00001. PMID 19078466
- [Background] Hanten WP, Olson SL, Butts NL, Nowicki AL. Effectiveness of a home program of ischemic pressure followed by sustained stretch for treatment of myofascial trigger points. Phys Ther. 2000 Oct;80(10):997-1003. PMID 11002435
- [Background] Desai MJ, Bean MC, Heckman TW, Jayaseelan D, Moats N, Nava A. Treatment of myofascial pain. Pain Manag. 2013 Jan;3(1):67-79. doi: 10.2217/pmt.12.78. PMID 24645933
- [Background] Lavelle ED, Lavelle W, Smith HS. Myofascial trigger points. Anesthesiol Clin. 2007 Dec;25(4):841-51, vii-iii. doi: 10.1016/j.anclin.2007.07.003. PMID 18054148
- [Background] Simons DG. Review of enigmatic MTrPs as a common cause of enigmatic musculoskeletal pain and dysfunction. J Electromyogr Kinesiol. 2004 Feb;14(1):95-107. doi: 10.1016/j.jelekin.2003.09.018. PMID 14759755
- [Background] Stifano G, Colantuono S, Carusi V, La Marra F, Marra A, Granata M. A case of tension-type headache in fibromyalgia. J Headache Pain. 2010 Aug;11(4):367-8. doi: 10.1007/s10194-010-0218-z. Epub 2010 May 9. No abstract available. PMID 20454992